CLINICAL TRIAL: NCT01562405
Title: Phase 1, Multicenter, Open-label, Dose-escalation Study of Sotatercept (ACE-011) in Combination With Lenalidomide or Pomalidomide and Dexamethasone in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Sotatercept (ACE-011) With Lenalidomide or Pomalidomide and Dexamethasone in Relapsed/Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Multiple Myeloma Research Consortium (Network)
Responsible Party: Principal Investigator, Andrew Yee, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-318
Record Dates: First submitted 2012-01-08; First posted 2012-03-23 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — ACE-011; Lenalidomide; Dexamethasone; Calcium Dobesilate; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACE-011 (sotatercept) (Experimental): ACE-011, Lenalidomide or pomalidomide, Dexamethasone
  Interventions: Drug: ACE-011; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Pomalidomide

INTERVENTIONS:
Drug: ACE-011 — Injection every 28 days, dose escalation levels from 15-45 mg
  Other Names: Sotatercept
Drug: Lenalidomide — 15 to 25 mg days 1-21, given orally
  Other Names: Revlimid
Drug: Dexamethasone — 40 mg days 1,8,15,22; given orally
  Other Names: Decadron
Drug: Pomalidomide — Pomalidomide 4 mg daily on days 1-21
  Other Names: Pomalyst

SUMMARY:
It is possible that the combination of lenalidomide, dexamethasone and ACE 011 may reduce or prevent the growth of cancer cells along with improving anemia and bone lesions that sometimes occur in people with multiple myeloma.

This current study is the first study combining ACE 011 with lenalidomide. In this research study, the investigators are looking for the highest dose of ACE 011 that can be given with lenalidomide and dexamethasone. The investigators will also begin to collect information about the effect of the combination of ACE 011, lenalidomide and dexamethasone on multiple myeloma.

DETAILED DESCRIPTION:
After the screening procedures confirm that you are eligible to participate in the research study:

Assignment to dose level of study treatment Since we are looking for the highest dose of the ACE 011 combined with lenalidomide that can be administered safely without severe or unmanageable side effects in participants that have multiple myeloma, not everyone who participates in this research study will receive the same dose of these drugs. The dose you get will depend on the number of participants who have been enrolled in the study before you and how well they have tolerated their doses.

Study treatment Study treatment will be given in 28 day cycles.

* ACE-011 will be given as an injection under the skin, Day 1 of each cycle (every 28 days). You will receive each injection at the clinic.
* Lenalidomide will be taken by mouth: once daily days 1 21, followed by a 7 day rest period during which no lenalidomide will be taken.
* Dexamethasone will be taken by mouth once per week (days 1, 8, 15 and 22) of each cycle.

You will be given drug diaries to record the doses of lenalidomide and dexamethasone taken. The study staff will tell you how to complete the diaries

ELIGIBILITY:
Inclusion Criteria:

* Monoclonal plasma cells in the bone marrow > 10% and/or presence of a biopsy-proven plasmacytoma
* Monoclonal protein present in the serum and/or urine
* Patient must have received at least 1 line of prior systemic therapy for the treatment of multiple myeloma. A line of treatment is sequential treatment without interruption for response and subsequent progression
* For participants treated with local radiotherapy with or without concomitant exposure to steroids, for pain control or management of cord/nerve root compression, two weeks must have lapsed since last date of radiotherapy, which is recommended to be a limited field. Participants who require concurrent radiotherapy should have entry to the protocol deferred until the radiotherapy is completed and two weeks have passed since the last date of therapy.
* ECOG performance status of zero to two unless decline is due to bony disease
* Not pregnant or breastfeeding

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants may not have received treatment with another investigational drug or device within 28 days prior to Day 1, or if the half life of the previous product is known, within 5 times the half life prior to dosing, whichever may be longer
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ACE 011, Lenalidomide or Dexamethasone
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* History of major surgery within 30 days prior to trial initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-05; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of ACE-011 | 2 years
  Identify the maximum tolerated dose of ACE-011 given in combination with lenalidomide and dexamethasone in subjects with relapsed multiple myeloma

SECONDARY OUTCOMES:
Efficacy of ACE-011 | 2 years
  * Objective response according to the International Myeloma Working Group Uniform Response Criteria
  * Duration of response
  * Time to progression
  * Progression-free survival
Safety of ACE-011 | 2 years
  * Adverse events profile
  * Toxicity profile as per NCI CTCAE v4.0
Pharmacodynamic measures | 2 years
  -Activin levels
Pharmacodynamic markers | 2 years
  Markers of bone turnover

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Yee, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Scullen T, Santo L, Vallet S, Fulciniti M, Eda H, Cirstea D, Patel K, Nemani N, Yee A, Mahindra A, Raje N. Lenalidomide in combination with an activin A-neutralizing antibody: preclinical rationale for a novel anti-myeloma strategy. Leukemia. 2013 Aug;27(8):1715-21. doi: 10.1038/leu.2013.50. Epub 2013 Feb 18. PMID 23417027